A comparative analysis between College Park Sidekick Feet and conventional stubby prosthesis.

NCT02921295

Sep 27, 2016

## Statistical Plan

A two-way analysis of variance (ANOVA) as a between subject variable and within subject variable will be used to analyze the dependent variable, completion time in seconds. A secondary analysis will observe additional dependent variables: cadence, velocity, step length, stride length, and pelvic girdle angles. The independent variables being analyzed include stubby feet compared with the Sidekicks and a level surface compared to gravel. The two-way ANOVA is used to determine whether there are any significant differences between the mean values of the independent groups. If a significant difference is detected an unpaired t-test will be implemented to determine if statistical significance exists. A probability value of 0.05 will be set at the level of statistical significance. Statistical analysis will be performed on SPSS software. The balance confidence scale and RPE scale will be compared across independent variables.